CLINICAL TRIAL: NCT07113522
Title: A Phase 2, Multi-Center, Platform Study to Evaluate the Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics With Multiple Therapies in Participants With Active Crohn's Disease or Active Ulcerative Colitis (ASCEND-IBD)
Brief Title: A Phase 2 Study to Evaluate Therapies for Inflammatory Bowel Disease
Acronym: ASCEND-IBD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mirador Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MT-100-201
Record Dates: First submitted 2025-07-15; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Inflammatory Bowel Disease (IBD); Ulcerative Colitis (UC); Crohn's Disease
Keywords: Inflammatory Bowel Diseases; ASCEND-IBD; Ulcerative Colitis; UC; CD; Crohn's Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Prospective Observer-Blinded Endpoint
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention Specific Appendix- Crohn's Disease (Experimental): Participants will receive MT-501
  Interventions: Drug: MT-501
- Intervention Specific Appendix- Ulcerative Colitis (Experimental): Participants will receive MT-501
  Interventions: Drug: MT-501

INTERVENTIONS:
Drug: MT-501 — MT-501 Tablets

SUMMARY:
This is a Phase 2, multicenter, platform study in adult participants with IBD (moderately to severely active Crohn's Disease or Ulcerative Colitis). The primary goal of this study is to assess the safety and efficacy of multiple investigational drugs.

DETAILED DESCRIPTION:
The purpose of this platform study is to assess the safety, efficacy, pharmacokinetics (PK), and pharmacodynamics (PD) to evaluate multiple oral or parenteral experimental therapies for moderately to severely active Crohn's Disease or Ulcerative Colitis.

ELIGIBILITY:
Inclusion Criteria-Crohn's Disease:

* Diagnosis of Crohn's Disease (CD), as confirmed by endoscopy and histopathology
* Moderately to severely active CD as defined by Clinical Disease Activity Index (CDAI) and Simple Endoscopic Score (SES-CD)
* Meets drug stabilization requirements

Inclusion Criteria-Ulcerative Colitis:

* Diagnosis of Ulcerative Colitis (UC), as confirmed by endoscopy and histopathology
* Moderately to severely active UC as defined by a 3-component MMCS
* Meets drug stabilization requirements

Exclusion Criteria-Crohn's Disease:

* Diagnosis of indeterminate colitis
* Suspected or diagnosed intra-abdominal or perianal abscess at Screening
* Previous small bowel resection with combined resected length of > 100 cm or previous colonic resection of > 2 segments
* CD isolated to the stomach, duodenum, jejunum, or perianal region, without colonic and/or ileal involvement

Exclusion Criteria-Ulcerative Colitis:

* Current evidence or within recent history (within last 6 months) of fulminant colitis, toxic megacolon, or bowel perforation
* Current stoma or impending need for colostomy or ileostomy
* Received IV corticosteroids within 14 days prior to Screening or during the Screening Phase
* Previous total proctocolectomy or subtotal colectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-05-07 (Estimated)

PRIMARY OUTCOMES:
Assess the proportion of participants reporting treatment emergent adverse events (TEAEs), serious adverse events (SAEs), adverse events (AEs) leading to discontinuation, and markedly abnormal laboratory values | Up to 13 weeks
Assess the Proportion of Participants with Endoscopic Response (CD) | 13 weeks
  Endoscopic response as assessed by SES-CD score.
Assess the Proportion of Participants Endoscopic Improvement (UC) | 12 weeks
  Endoscopic improvement as assessed by MES.
Assess the Proportion of Participants with Clinical Remission (CD) | 13 weeks
  Clinical remission as assessed by CDAI score.
Assess the Proportion of Participants with Clinical Remission (UC) | 12 weeks
  Clinical remission as assessed by endoscopy, rectal bleeding and stool frequency.

SECONDARY OUTCOMES:
Assess the Proportion of Participants with Clinical Remission (CD) | 13 weeks
  CD: Clinical remission as assessed by CDAI score.
Assess the Proportion of Participants with Clinical Remission (UC) | 12 weeks
  Clinical remission as assessed by endoscopy, rectal bleeding, and stool frequency.
Assess the Proportion of Participants with Symptomatic Remission (CD and UC) | Up to 13 weeks
  Symptomatic remission as assessed by patient reported outcomes.
Assess the Proportion of Participants with Clinical Response (CD) | 13 weeks
  CD: Clinical response as assessed by CDAI score.
Assess the Proportion of Participants with Clinical Response (UC) | 12 weeks
  UC: Clinical response as assessed by MMCS.
Assess the Proportion of Participants with Endoscopic and Clinical Response (CD Only) | 13 weeks
  Endoscopy as assessed by SES-CD and clinical response as assessed by CDAI score.
Assess the Proportion of Participants with Histologic Response (UC Only) | 12 weeks
  Histologic response as assessed by the RHI.
Assess the Proportion of Participants with Histologic Remission (UC only) | 12 weeks
  Histologic remission as assessed by the RHI.
Assess the Proportion of Participants with Histologic-Endoscopic Mucosal Improvement (UC only) | 12 weeks
  Histologic-endoscopic mucosal improvement as assessed by the Geboes score and MES.
Characterize the Change in Endoscopy Score (CD) | 13 weeks
  CD: Endoscopy score as assessed by SES-CD.
Characterize the Change in Endoscopy Score (UC) | 12 weeks
  Endoscopy score as assessed by MES.
Characterize the Change in Histology Score (CD) | 13 weeks
  Histology as assessed by GHAS and RHI.
Characterize the Change in Histology Score (UC) | 12 weeks
  Histology as assessed by Geobes, RHI and NHI
Asses the Pharmacokinetics (PK) (e.g., Trough Concentration [Ctrough]) of Investigational Drug | Up to 13 weeks

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Mirador Therapeutics Selected Site, Little Rock, Arkansas
  - Mirador Therapeutics Selected Site, Miami, Florida
  - Mirador Therapeutics Selected Site, Orlando, Florida
  - Mirador Therapeutics Selected Site, Snellville, Georgia
  - Mirador Therapeutics Selected Site, Glenview, Illinois
  - Mirador Therapeutics Selected Site, Shreveport, Louisiana
  - Mirador Therapeutics Selected Site, Liberty, Missouri
  - Mirador Therapeutics Selected Site, Rochester, New York
  - Mirador Therapeutics Selected Site, Greenville, South Carolina
  - Mirador Therapeutics Selected Site, Cordova, Tennessee
  - Mirador Therapeutics Selected Site, Dallas, Texas
  - Mirador Therapeutics Selected Site, Georgetown, Texas
  - Mirador Therapeutics Selected Site, Lubbock, Texas
  - Mirador Therapeutics Selected Site, Southlake, Texas
  - Mirador Therapeutics Selected Site, Tyler, Texas
  - Mirador Therapeutics Selected Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No